CLINICAL TRIAL: NCT04788940
Title: Clinical Implication of Cardiac Magnetic Resonance Imaging for Patients With Acute Myocardial Infarction: Prospective Observational Study
Brief Title: Clinical Implication CMR in AMI Registry
Acronym: CMR-AMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Young Bin Song, Professor, Samsung Medical Center
Other Study IDs: CMR-AMI 2021
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Acute Myocardial Infarction
Keywords: Percutaneous Coronary Intervention; Acute Myocardial Infarction; Cardiac Magnetic Resonance Imaging
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AMI patients treated with PCI: Acute myocardial infarction patients who underwent percutaneous coronary intervention and cardiac magnetic resonance imaging
  Interventions: Procedure: Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention — Patients with AMI who underwent PCI and CMR at index hospitalization and 6-month follow-up

SUMMARY:
1. To evaluate the clinical implication of cardiac magnetic resonance imaging in patients with acute myocardial infarction
2. To determine factors affecting the 6-month remodeling index assessed by cardiac magnetic resonance imaging

DETAILED DESCRIPTION:
To date, advances in medical treatment and reperfusion therapy led to markedly decreased morbidity and mortality rate in patients with acute myocardial infarction (AMI). Nevertheless, there is a deterioration of left ventricular systolic function or development of heart failure in 40-50% of surviving patients with AMI after the percutaneous coronary intervention (PCI), and it is related to infarct size at the index procedure. Conventional methods of measuring the infarct size included electrocardiogram, peak cardiac enzyme, and echocardiography, but these do not indicate the exact irreversible tissue damage and only suggest indirect parameters. However, cardiac magnetic resonance imaging (CMR) provides information on infarct size, microvascular obstruction, transmurality, and salvage index, and discriminative function between viable and non-viable myocardium with high spatial resolution. Also, magnetic resonance imaging is used as a gold standard for the evaluation of the myocardial remodeling index. However, it is not well known in which patients occur adverse remodeling for the myocardium and in which patients occur reverse remodeling. Therefore, the investigators sought to evaluate the clinical implication of CMR and to determine factors affecting the 6-month remodeling index assessed by cardiac magnetic resonance imaging through the current registry.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed as type 1 myocardial infarction the presence of acute myocardial injury detected by abnormal cardiac biomarkers in the setting of evidence of acute myocardial ischemia.

Exclusion Criteria:

* Patients who cannot perform cardiac magnetic resonance imaging
* Target vessel is not suitable for coronary intervention

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: About 500 patients with acute myocardial infarction and who underwent PCI.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in proportion of adverse/reverse remodeling at 6 months | at 6-month follow-up
  Remodeling index assessed by baseline and follow-up CMR

SECONDARY OUTCOMES:
Infarct size | 72 hours after the index procedure
  Infarct size assessed by baseline CMR
Myocardial salvage index | 72 hours after the index procedure
  Myocardial salvage index assessed by baseline CMR
Microvascular obstruction | 72 hours after the index procedure
  Microvascular obstruction assessed by baseline CMR
Hemorrhagic infarct | 72 hours after the index procedure
  Hemorrhagic infarct assessed by baseline CMR
Transmurality | 72 hours after the index procedure
  Transmurality assessed by baseline CMR
Peak cardiac enzyme | 72 hours after the index procedure
  Peak cardiac enzyme at index hospitalization
TIMI flow | Immediate after the index procedure
  TIMI flow grade after culprit vessel PCI
Changes of LVEDV on CMR | at 6-month follow-up
  ∆left ventricular end diastolic volume assessed by baseline and follow-up CMR
Changes of LVESV on CMR | at 6-month follow-up
  ∆left ventricular end systolic volume assessed by baseline and follow-up CMR
6-month Infarct size | at 6-month follow-up
  Infarct size assessed by 6-month CMR
6-month myocardial salvage index | at 6-month follow-up
  myocardial salvage index assessed by 6-month CMR
6-month microvascular obstruction | at 6-month follow-up
  6-month microvascular obstruction assessed by 6-month CMR
6-month hemorrhagic infarct | at 6-month follow-up
  6-month hemorrhagic infarct assessed by 6-month CMR
Changes of LVEDV on echocardiography | at 6-month follow-up
  ∆left ventricular end diastolic volume assessed by baseline and follow-up echocardiography
Changes of LVESV on echocardiography | at 6-month follow-up
  ∆left ventricular end systolic volume assessed by baseline and follow-up echocardiography
Changes of LVEF on echocardiography | at 6-month follow-up
  ∆left ventricular ejection fraction assessed by baseline and follow-up echocardiography
Cardiac death or heart failure readmission | 1-year after last patient enrollment
  Cardiac death or heart failure readmission during follow-up
All-cause death or heart failure readmission | 1-year after last patient enrollment
  All-cause death or heart failure readmission during follow-up
Target lesion failure | 1-year after last patient enrollment
  a composite of cardiac death, myocardial infarction, clinically driven target lesion revascularization
target vessel failure | 1-year after last patient enrollment
  a composite of cardiac death, myocardial infarction, clinically driven target vessel revascularization
All-cause death | 1-year after last patient enrollment
  Rate of all-cause death during follow-up
Cardiac death | 1-year after last patient enrollment
  Rate of cardiac death during follow-up
Myocardial infarction | 1-year after last patient enrollment
  Myocardial infarction during follow-up
Target vessel myocardial infarction | 1-year after last patient enrollment
  Rate of Target vessel myocardial infarction during follow-up
Target lesion revascularization | 1-year after last patient enrollment
  Rate of target lesion revascularization during follow-up
Target vessel revascularization | 1-year after last patient enrollment
  Rate of target vessel revascularization during follow-up
Heart failure readmission | 1-year after last patient enrollment
  Rate of heart failure readmission during follow-up
Any readmission | 1-year after last patient enrollment
  Rate of any readmission during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Young Bin Song, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea